CLINICAL TRIAL: NCT07343011
Title: Conjunctival Transpositional Pterygium Surgery: A Prospective Single-Arm Interventional Study
Brief Title: Conjunctival Transpositional Surgery for Primary Pterygium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammed Arish, Associate professor of ophthalmology, Zahedan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.ZAUMS.REC.1404.238
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pterygium of the Conjunctiva and Cornea
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pterygium patients (Experimental)
  Interventions: Procedure: Conjunctival Transpositional Pterygium Surgery

INTERVENTIONS:
Procedure: Conjunctival Transpositional Pterygium Surgery — A conjunctival incision was created at the upper and lower limbus to allow adequate tissue mobilization. The pterygium tissue is dissected off the corneal surface without complete excision or creation of a bare sclera defect. The fibrovascular tissue is mobilized and transposed inferiorly within the subconjunctival plane and secured with absorbable sutures. Tenon's tissue is preserved, and no adjunctive therapy is used.

SUMMARY:
This prospective single-arm interventional study evaluates the recurrence rate and functional outcomes following conjunctival transpositional pterygium surgery without bare sclera formation. The technique involves mobilization and transposition of the pterygium tissue while preserving Tenon's layer and avoiding adjunctive therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Primary pterygium involving the cornea
* Ability to provide informed consent

Exclusion Criteria:

* Recurrent pterygium
* Previous ocular surface surgery
* Active ocular infection or inflammation
* Severe ocular surface disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Pterygium Recurrence | 12 months
  Recurrence is defined as fibrovascular regrowth toward the cornea or surgical failure.

SECONDARY OUTCOMES:
Visual Acuity | 12 months
  Change in visual acuity measured in logMAR units.
Refractive Astigmatism | 12 months
  Change in refractive astigmatism measured as cylindrical power in diopters.

CONTACTS AND LOCATIONS:
Locations (1):
- Alzahra Eye Hospital, Zahedan University of Medical Sciences, Zahedan, Sistan and Balochistan, Iran

IPD SHARING:
Plan to Share IPD: Undecided